CLINICAL TRIAL: NCT01566838
Title: A Randomized Controlled Trial of Continuous Subpleural Infusion of Bupivacaine After Thoracoscopy
Brief Title: Continuous Subpleural Infusion of Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120104onq
Record Dates: First submitted 2012-02-21; First posted 2012-03-29 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain
Keywords: Visual analog pain score; Length of stay; Hospital Cost; Subpleural pain catheter; Bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-q pump (Active Comparator): Patients in this arm will receive the standard acute pain management regimen during hospital admission and will be sent home after discharge with a subpleural pain catheter and instructions for removal when pump is empty (around 5 days time). The catheter will contain an infusion of 0.125% bupivacaine. The single lumen pain catheter is infused by a self deflating pump filled to 335ml, which delivers the infusate at a rate of 4ml/h. Pumps are expected to be empty in 4 to 5 days.
  Interventions: Drug: Subpleural pain catheter with infusion of 0.125% bupivacaine
- Standard of care (Active Comparator): Patients in this arm will not receive a pain catheter in addition to the standard of care for pain management. Standard of care will consist of a standard balanced anesthetic consisting of midazolam 0.01-0.03mg/kg, induced with propofol (1-2mg/kg) or etomidate, fentanyl (1-2 mcg/kg) and rocuronium (0.1mg/kg) and maintained on a potent inhalation agent (sevoflurane 1.5%-2.5%) during procedures. Prior to emergence from anesthesia, patients will receive ketorolac 30mg IV once, neuromuscular reversal agents, and an antiemetic (ondansetron 4mg). Patients will also be given additional narcotics (fentanyl) upon emergence, as needed, to facilitate patient comfort and extubation.
  The ASA guidelines for acute pain management in the perioperative period will also be provided. Patients shall receive 1,000 mg of acetaminophen orally every 6 hours, scheduled for 5 days. Other drugs will be given on as needed basis (PRN) to maintain an analog pain scale of ≤ 3.
  Interventions: Drug: Standard acute pain management

INTERVENTIONS:
Drug: Subpleural pain catheter with infusion of 0.125% bupivacaine — Patients in this arm will be provided with a subpleural pain catheter and instructions for removal when pump is empty (around 5 days time). The catheter will contain an infusion of 0.125% bupivacaine. The single lumen pain catheter is infused by a self deflating pump filled to 335ml, which delivers the infusate at a rate of 4ml/h. Pumps are expected to be empty in 4 to 5 days.
  Other Names: On-q pump
  Arms: On-q pump
Drug: Standard acute pain management — A standard balanced anesthetic consisting of midazolam 0.01-0.03mg/kg, induced with propofol (1-2mg/kg) or etomidate, fentanyl (1-2 mcg/kg) and rocuronium (0.1mg/kg) and a potent inhalation agent (sevoflurane 1.5%-2.5%) during procedures.
  Prior to emergence from anesthesia, patients will receive ketorolac 30mg IV, neuromuscular reversal agents, and ondansetron 4mg. Fentanyl will be given, as needed, to facilitate patient comfort and extubation.
  The ASA guidelines for acute pain management in the perioperative period will be followed. Patients shall receive 1,000 mg of acetaminophen orally every 6 hours, scheduled for 5 days. Other drugs will be given on as needed basis (PRN) to maintain an analog pain scale of ≤ 3.
  Arms: Standard of care

SUMMARY:
Rationale: For the past 3 years the investigators have routinely used an axial subpleural tunneling technique that del

Study Design: All patients over the age of 18 having an isolated thoracoscopic procedure performed at Inova Fairfax Hospital for therapeutic or diagnostics purposes will be screened. Patients will be excluded if they have: previous ipsilateral thoracic surgery, need for operative pleurectomy or pleurodesis, chronic use of pain medication, sedatives or hypnotics, drug allergies, liver dysfunction, renal dysfunction, history of peptic ulcerative disease, sleep apnea in need of Bipap, severe chronic obstructive pulmonary disease (COPD), inability to consent, or are pregnant. All patients included will be screened, consented, and operated on by the one year anniversary of institutional review board (IRB) approval.

Study Methodology: Eighty-six consented patients will be randomized into the study arm (use of a pain catheter with 0.125% bupivacaine) or the standard of care group (no pain catheter). The primary outcome is the use of narcotic pain medication post-operatively, compared between study groups. Secondary outcomes will include postoperative pain scores, hospital and length of stay.

The On-Q pump delivers local anesthetic to the intercostal space, without leakage elsewhere, creating a functional multi level rib block. Despite positive subjective results, objective data is lacking. The investigators have also noted that some patients develop an annoying short term paresthesia that has been minimized by using lower anesthetic concentrations than described in other publications.

Objectives: To evaluate visual analog pain scores post-operatively up to 30 days post-operative, and to determine any association between pain management and length of stay.

Study Type: A prospective randomized 2-arm study will be performed. Statistical Methodology: Total amount of narcotic pain medication administered through postoperative day 7, will be compared between the study groups using student's t-tests and Wilcoxon rank-sum tests. Secondary outcomes, overall sum of pain scores through postoperative day 7, then at day 30 post-operatively, hospital length of stay, and overall hospital cost, will also be compared among study groups using student's t-tests and Wilcoxon rank-sum tests.

DETAILED DESCRIPTION:
Video-Assisted Thoracic Surgery (VATS) has been shown to hasten patient recovery by attenuating the physiologic stress of surgery and decreasing post-operative pain. Despite this approach, incisions in the chest are proportionally more painful than in other parts of the body, and most patients require some form of narcotic pain medication.

Multiple strategies for post-operative pain control have been attempted in thoracic surgery with no obvious superiority of one versus another. Pain catheters have been increasingly used over the past decade in different surgical procedures in order to minimize incisional pain for the first 3 to 7 days after an operation. The published literature is equivocal as to the efficacy of such approach following thoracic surgery with most recent series reporting no benefit in the use of these catheters. Of utmost importance is the placement techniques described thus far, which in our opinion, have been suboptimal.

In order for a pain catheter to work, the infused local anesthetic has to constantly bathe the nerve in question thus preventing painful stimuli from being transmitted. It is hard to dispute the ability of local anesthetic to block pain conduction. Consequently, the success of the intervention is directly dependent on the placement technique to achieve such goal, hence the rationale for our study.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age
* Isolated thoracoscopic procedure for therapeutic or diagnostic purposes

Exclusion Criteria:

* Previous ipsilateral thoracic surgery
* Need for operative pleurectomy or pleurodesis
* Chronic use of pain medication (narcotics or NSAIDS), sedatives or hypnotics
* Allergies to bupivacaine or other local anesthetics, narcotics, NSAIDs or acetaminophen
* Liver dysfunction (INR > 1.5, albumin < 2.8g/dl, bilirubin > 2mg/dl)
* Renal dysfunction (eGFR < 60ml/min/1.73m2)
* History of peptic ulcerative disease
* Sleep apnea in need of Bipap
* Severe COPD requiring continuous oxygen supplementation
* Inability to consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Fortes, MD, Principal Investigator — Cardiac, Vascular, & Thoracic Surgery Associates
Locations (1):
- Inova Fairfax Hospital, Falls Church, Virginia, United States

REFERENCES:
- [Background] Whitson BA, Groth SS, Duval SJ, Swanson SJ, Maddaus MA. Surgery for early-stage non-small cell lung cancer: a systematic review of the video-assisted thoracoscopic surgery versus thoracotomy approaches to lobectomy. Ann Thorac Surg. 2008 Dec;86(6):2008-16; discussion 2016-8. doi: 10.1016/j.athoracsur.2008.07.009. PMID 19022040
- [Background] Allen MS, Halgren L, Nichols FC 3rd, Cassivi SD, Harmsen WS, Wigle DA, Shen KR, Deschamps C. A randomized controlled trial of bupivacaine through intracostal catheters for pain management after thoracotomy. Ann Thorac Surg. 2009 Sep;88(3):903-10. doi: 10.1016/j.athoracsur.2009.04.139. PMID 19699918
- [Background] Chan VW, Chung F, Cheng DC, Seyone C, Chung A, Kirby TJ. Analgesic and pulmonary effects of continuous intercostal nerve block following thoracotomy. Can J Anaesth. 1991 Sep;38(6):733-9. doi: 10.1007/BF03008451. PMID 1914056
- [Background] Gurvich EB, Gladkova EV. [The results and outlook of a clinico-epidemiological study of the problem of the carcinogenic hazard in industry]. Gig Tr Prof Zabol. 1992;(7):17-20. Russian. PMID 1296910
- [Background] Kaiser AM, Zollinger A, De Lorenzi D, Largiader F, Weder W. Prospective, randomized comparison of extrapleural versus epidural analgesia for postthoracotomy pain. Ann Thorac Surg. 1998 Aug;66(2):367-72. doi: 10.1016/s0003-4975(98)00448-2. PMID 9725371
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2004 Jun;100(6):1573-81. doi: 10.1097/00000542-200406000-00033. No abstract available. PMID 15166580

RESULTS

PARTICIPANT FLOW:
Groups:
- On-q Pump: Patients in this arm will receive the standard acute pain management regimen during hospital admission and will be sent home after discharge with a subpleural pain catheter and instructions for removal when pump is empty (around 5 days time). The catheter will contain an infusion of 0.125% bupivacaine. The single lumen pain catheter is infused by a self deflating pump filled to 335ml, which delivers the infusate at a rate of 4ml/h. Three patients did not have follow-up data for the study and were therefore excluded from analysis
  Subpleural pain catheter with infusion of 0.125% bupivacaine: Patients in this arm will be provided with a subpleural pain catheter and instructions for removal when pump is empty (around 5 days time). The catheter will contain an infusion of 0.125% bupivacaine. The single lumen pain catheter is infused by a self deflating pump filled to 335ml, which delivers the infusate at a rate of 4ml/h. Pumps are expected to be empty in 4 to 5 days.
- Standard of Care: Patients in this arm will not receive a pain catheter in addition to the standard of care for pain management. Standard of care will consist of a standard balanced anesthetic consisting of midazolam 0.01-0.03mg/kg, induced with propofol (1-2mg/kg) or etomidate, fentanyl (1-2 mcg/kg) and rocuronium (0.1mg/kg) and maintained on a potent inhalation agent (sevoflurane 1.5%-2.5%) during procedures. Prior to emergence from anesthesia, patients will receive ketorolac 30mg IV once, neuromuscular reversal agents, and an antiemetic (ondansetron 4mg). Patients will be given additional narcotics (fentanyl) upon emergence, as needed, to facilitate patient comfort and extubation.
  The ASA guidelines for acute pain management in the perioperative period will also be provided. Patients shall receive 1,000 mg of acetaminophen orally every 6 hours, scheduled for 5 days. Other drugs will be given on as needed basis (PRN) to maintain an analog pain scale of ≤ 3.
  Standard acute pain management
Period: Overall Study
Arm/Group | On-q Pump | Standard of Care
Started | 41 | 42
Completed | 38 | 42
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-q Pump | Standard of Care | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.4) | 62.9 (12.1) | 62.95 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 20 | 21 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 34 | 35 | 69
  Other | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 41 | 42 | 83
Surgical Procedure Performed [Number; unit: participants]
  Lobectomy | 23 | 20 | 43
  Wedge | 18 | 16 | 34
  Other | 0 | 6 | 6
Diagnosis [Number; unit: participants]
  Cancer | 30 | 27 | 57
  Interstitial Lung Disease | 7 | 12 | 19
  Other | 4 | 3 | 7
Side [Number; unit: participants]
  Left | 11 | 12 | 23
  Right | 30 | 29 | 59
  Unspecified | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without 30-Day Pain Medication Usage
Description: The primary outcome will measure narcotics usage from post-operative day 1 through post-operative day 30.
Time Frame: Postoperative day 1 through postoperative day 30
Population: 30-day pain medication usage
Measure: Number; unit: participants
Arm/Group | On-q Pump | Standard of Care
Number analyzed (Participants) | 38 | 42
participants
  Yes | 8 | 6
  No | 30 | 36

2. Secondary Outcome: 7-day Paresthesia
Description: Participants experiencing parasthesia (a tingling or pricking sensation usually caused by pressure or damage to nerves) through postoperative day 7
Time Frame: Postoperative day 1 through day 7
Population: 7-day paresthesia
Measure: Number; unit: participants
Arm/Group | On-q Pump | Standard of Care
Number analyzed (Participants) | 38 | 42
participants
  Yes | 3 | 1
  No | 25 | 25
  Unknown | 10 | 16

3. Secondary Outcome: Length of Stay
Description: Hospital length of stay for this operation will be recorded and analyzed for each arm of the study.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Population: In-hospital length of stay (days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | On-q Pump | Standard of Care
Number analyzed (Participants) | 38 | 42
days | 1 [0 to 1] | 1 [0 to 1]

4. Secondary Outcome: 30-day Incidence of Parasthesia
Description: 30-day incidence of paresthesia (tingling or pricking sensation, usually caused by pressure or nerve damage)
Time Frame: 30 days
Population: 30-day incidence of paresthesia
Measure: Number; unit: participants
Arm/Group | On-q Pump | Standard of Care
Number analyzed (Participants) | 38 | 42
participants
  Yes | 13 | 15
  No | 25 | 27

5. Secondary Outcome: Return to Work
Description: Returned to work in 30 days?
Time Frame: 30 days
Population: 30 day return to work
Measure: Number; unit: participants
Arm/Group | On-q Pump | Standard of Care
Number analyzed (Participants) | 38 | 42
participants
  Yes | 18 | 20
  No | 3 | 3
  Not currently working | 17 | 19

6. Secondary Outcome: Resumed Physical Activity
Description: Did the patient resume physical activity.
Time Frame: 30 days
Population: Resuming of physical activity
Measure: Number; unit: participants
Arm/Group | On-q Pump | Standard of Care
Number analyzed (Participants) | 38 | 42
participants
  Yes | 37 | 37
  No | 1 | 5

ADVERSE EVENTS:
Arm/Group | On-q Pump | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/42

LIMITATIONS AND CAVEATS:
This study limited by a low power and reliance on patient self-reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No